CLINICAL TRIAL: NCT06198751
Title: A Phase 2, Randomized, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of TQB2102 for Injection for Neoadjuvant Treatment of Breast Cancer With Positive HER2 Expression
Brief Title: A Study of Neoadjuvant Treatment With TQB2102 for Injection for Human Epidermal Growth Factor Receptor 2 (HER2) Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-II-01
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 mg/kg of TQB2102 for injection (Experimental): 6 mg/kg TQB2102, Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle, for 6 or 8 cycles.
  Interventions: Drug: 6.0 mg/kg of TQB2102 for injection
- 7.5 mg/kg of TQB2102 for injection (Experimental): 7.5 mg/kg TQB2102, Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle, for 6 or 8 cycles.
  Interventions: Drug: 7.5 mg/kg of TQB2102 for injection

INTERVENTIONS:
Drug: 6.0 mg/kg of TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC), 6.0 mg/kg.
  Arms: 6 mg/kg of TQB2102 for injection
Drug: 7.5 mg/kg of TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC), 7.5 mg/kg.
  Arms: 7.5 mg/kg of TQB2102 for injection

SUMMARY:
To evaluate the efficacy and safety of neoadjuvant treatment with TQB2102 for injection in patients with Her2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study and sign informed consent;
* Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1; expected survival of more than 3 months;
* Histologically confirmed invasive breast cancer, no history of any systemic anti-tumor therapy for breast cancer;
* Confirmed as HER2 positive;
* Clinical stage at the time of visit is T0-4, N1-3, M0 or T2-4, N0, M0;
* Agree to undergo breast cancer surgery when reaching the surgical criteria after neoadjuvant therapy;
* Major organ functions are good, meeting certain criteria;
* Agree to use contraception during the study and within 6 months after the study ends; female patients must have a negative serum pregnancy test within 7 days before enrollment and must be non-lactating.

Exclusion Criteria:

* IV stage metastatic breast cancer or deemed unable to achieve curative surgical resection through neoadjuvant therapy by other investigators.
* Bilateral invasive breast cancer.
* Coexisting diseases and medical history:

  1. History of invasive breast cancer.
  2. Occurrence of any other malignant tumors within the last 3 years or current simultaneous presence.
  3. Underwent significant surgical treatment, incisional biopsy, or significant trauma within 28 days before the start of the study.
  4. Unhealed wounds or fractures.
  5. Ocular diseases deemed clinically significant by the investigator.
  6. Occurrence of arterial/deep venous thrombotic events within the last 6 months.
  7. History of substance abuse with inability to quit or individuals with mental disorders.
  8. ≥ Grade 2 myocardial ischemia or infarction, arrhythmias, or ≥ Grade 2 congestive heart failure.
  9. Uncontrolled ≥ CTCAE Grade 2 infection within 14 days before the start of the study.
  10. History of interstitial lung disease/pneumonia requiring intervention with steroid treatment, or current presence, or suspected interstitial lung disease/pneumonia during the screening period that cannot be ruled out by the investigator; individuals with pulmonary diseases deemed unsuitable for participation by the investigator.
* Tumor-related symptoms and treatment:

  1. Received surgery, chemotherapy, radiotherapy, or other anti-tumor therapy within 4 weeks before the start of the study.
  2. Received traditional Chinese medicine treatment with indications for anti-tumor effects within 2 weeks before the start of the study.
  3. Radiological evidence of tumor invasion into major vessels or judged by the investigator to be highly likely to invade major vessels during the subsequent study period, leading to fatal hemorrhage.
* Study treatment-related:

  1. Experienced severe hypersensitivity reactions after using monoclonal antibodies.
  2. Developed uncontrollable active autoimmune diseases within 2 weeks before the start of the study.
  3. Allergic to any component or excipient in any study drug.
* Participated in other clinical trials of anti-tumor drugs within 4 weeks before the start of the study.
* Deemed inappropriate for inclusion based on the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Total physiological complete response (tpCR) | Up to 12 months.
  The percentage of the patients where the primary breast lesion shows no residual infiltrating cancer and the regional lymph nodes are negative.

SECONDARY OUTCOMES:
Breast pathological complete (bpCR) response | Up to 12 months.
  The percentage of the patients where the primary breast lesion shows no residual infiltrating cancer.
Objective response rate (ORR) | Up to 12 months.
  The percentage of subjects achieving complete response (CR) or partial response (PR) as assessed by the investigator based on the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Event-free survival (EFS) | Up to 60 months.
  The time from the date of surgery completion to the first occurrence of the following events，including disease progression precluding surgery, ipsilateral or contralateral recurrence of invasive breast cancer, regional or distant recurrence of invasive breast cancer, a second primary malignancy in a non-breast site, and death for any reason.
Invasive Disease-free survival (IDFS) | Up to 60 months.
  The time from the date of surgery completion to the first occurrence of the following events，including ipsilateral or contralateral recurrence of invasive breast cancer, regional or distant recurrence of invasive breast cancer, a second primary malignancy in a non-breast site, and death for any reason.
The occurrence rate of all adverse events (AEs) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The occurrence of adverse events defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0)
The severity of all adverse events (AEs) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The severity of adverse events defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0).
Anti-drug antibody (ADA) | 1 hour Before infusion on Cycle 1 Day1, Cycle 2 Day1, Cycle 4 Day1, Cycle 6 Day1, Cycle 8 Day1, and 90 days after the end of the last infusion. Each cycle is 21 days.
  Incidence of anti-drug antibody (ADA)
Overall survival (OS) | Up to 60 months after study start
  The time from the date of surgery completion to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Harbin medical university cancer hospital, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Li JJ, Zhang WJ, Zeng XH, Zhang QY, Chen L, Wu J, Liu GY, Wang ZH, Hu XB, Hu YY, Li ZL, Shao ZM. Efficacy and Safety of Neoadjuvant TQB2102 in Locally Advanced or Early Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer: A Randomized, Open-Label, Multicenter, Phase II Trial. J Clin Oncol. 2026 Jan;44(1):20-30. doi: 10.1200/JCO-25-01153. Epub 2025 Nov 25. PMID 41289548